CLINICAL TRIAL: NCT00002091
Title: An Evaluation of Pentoxifylline in HIV-Positive Persons With Symptomatic HIV Infection and a Karnofsky Score > 40 Percent and < 100 Percent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 118A; 91-02
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-10

CONDITIONS: HIV Infections
Keywords: Pentoxifylline; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline

SUMMARY:
PRIMARY: To determine whether pentoxifylline changes the self-reported measures of quality of life status, using measures of scores from double-blinded drug withdrawal and drug restart periods.

SECONDARY: To measure the changes in monthly CD4 counts, fasting serum triglyceride levels, and weight; to assess the safety of pentoxifylline in HIV-infected persons.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Stable antiretroviral therapy.
* Maintenance medication for opportunistic infection.

Patients must have:

HIV positivity.

NOTE:

* Patients on an antiretroviral must have received it for at least 2 months and have no currently perceived need to change or add to the regimen for the next 3 months.

Prior Medication:

Allowed:

* Antiviral therapy (provided patient has been on such therapy for at least 2 months at study entry and dose is stable).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Evidence of active opportunistic infection or malignancy requiring high-dose systemic chemotherapy (only patients who are 30 days from a diagnosis of an opportunistic infection and on appropriate maintenance medication are allowed).
* Known significant intolerance or hypersensitivity to theophylline, theobromine (chocolate), or caffeine, for reasons other than dyspepsia.
* Inability to swallow tablets (gastric feeding tubes are allowed).
* Active bleeding disorder or major bleeding source, including peptic ulcer or gastritis.
* Any symptoms suggestive of concurrent illness that are not attributable to overall impairment by HIV or are not diagnosable based on the available evidence.
* Not willing to comply with visit schedule and study procedures.

Concurrent Medication:

Excluded:

* Concurrent use of the anticoagulant warfarin (Coumadin) and heparin.

Prior Medication:

Excluded:

* Treatment with biologic response modifiers (e.g., interferon, interleukin) within 14 days prior to study entry.

Prior Treatment:

Excluded:

* Major surgery within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (1):
- CRI of New England, Brookline, Massachusetts, United States

REFERENCES:
- [Background] Cohen CJ, Dezube BJ, Day JM, Andradas V, Gagnon S, Rieker PP. The impact of pentoxifylline on quality of life. Int Conf AIDS. 1994 Aug 7-12;10(1):213 (abstract no PB0283)